CLINICAL TRIAL: NCT00866866
Title: The Use of Oral N-Acetyl Cysteine for the Treatment of Chronic Sinonasal Symptoms: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: The Use of Oral N-Acetyl Cysteine for the Treatment of Chronic Sinonasal Symptoms
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Dr. B. Mechor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21571
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Last update posted 2009-03-23 (Estimated); Status verified 2009-03

CONDITIONS: Chronic Sinonasal Symptoms
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- N-Acetyl Cysteine (Experimental)
  Interventions: Drug: N-Acetyl Cysteine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-Acetyl Cysteine — 600 mg PO BID
  Arms: N-Acetyl Cysteine
Drug: Placebo — 1 tab PO BID
  Arms: Placebo

SUMMARY:
Chronic sinonasal symptoms (CSNS), such as coughing, throat clearing, nasal obstruction, crusting, dryness and discharge are extremely common in the general population. Although the physical symptoms are readily apparent, the psychosocial impact is often overlooked. Depression, anxiety, fear of social interaction, impaired personal relationships and decreased performance at work have all been associated with CSNS, often leading to multiple, frequent visits to the patient's primary care physician. A variety of clinical studies have shown that health-related quality of life (HRQoL) is significantly impaired in people with CSNS, with depressive symptoms being particularly common.

CSNS may be due, in part, to tenacious nasal and paranasal secretions. It is therefore conceivable that a mucolytic may thin these secretions and improve mucociliary clearance, thereby reducing CSNS. N-acetylcysteine (NAC) is the most widely used mucolytic agent, particularly in patients with cystic fibrosis (CF), and has been documented as the most effective of the mucokinetic agents. Our group wishes to examine the use of NAC as a treatment for CSNS by testing the hypothesis that oral NAC reduces symptoms of CSNS compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* one or more the following symptoms: nasal stuffiness, nasal dryness or crusting, nasal congestion, discolored nasal discharge, or thick nasal discharge, for four or more days a week in the preceding two weeks

Exclusion Criteria:

* poorly controlled asthma
* cystic fibrosis
* chronic obstructive pulmonary disease (COPD)
* severe coronary artery disease
* vasculopathy
* poorly controlled diabetes
* poorly controlled hypertension
* women who are breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-12 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Sinonasal Outcomes Test (SNOT) - 22 | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Warren Yunker, MD, PhD, Study Director — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada